CLINICAL TRIAL: NCT07370896
Title: The Alvarado Score in the Emergency Department of Hospitals in the Meta Department, Colombia. A Cross-sectional Study
Brief Title: Alvarado Score in the Meta Department
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU director, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2019_01_QX_Alvarado
Record Dates: First submitted 2025-12-15; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Appendicitis (Diagnosis); Acute Appendicitis
Keywords: Appendicitis; Acute Appendicitis; Diagnosis; Abdominal Pain; Acute Abdomen; Alvarado Score; Primary Care; Developing Countries; Colombia
MeSH Terms: conditions — Appendicitis; Disease; Abdominal Pain; Abdomen, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- City of the facility: Location of the facility
- Site of graduation: Physicians graduated in the local university

SUMMARY:
The project aims to determine the frequency of use of the Alvarado score among emergency department physicians at facilities in Villavicencio, Colombia. The information will be collected using a self-directed survey with items assessing awareness, compliance, and systematic recording of the Alvarado score among patients with abdominal pain and suspected acute appendicitis, as predictors of illness and severity.

DETAILED DESCRIPTION:
Introduction: Early detection of appendicitis in the emergency department is vital for prompt treatment and the prevention of complications. The Alvarado score is a diagnostic tool designed to predict the probability of appendicitis in adults. Publications about the use of the Alvarado score are limited. Understanding how frequently a predictive score is used is essential for promoting its adoption. This study aimed to assess the frequency with which emergency department physicians in healthcare facilities in the Meta Department use the Alvarado score.

Methodology: Between August 2019 and January 2020, a cross-sectional survey was conducted with physicians (N = 125) who voluntarily participated from five hospitals in the area.

ELIGIBILITY:
Inclusion Criteria:

* Graduated physician
* Working in the emergency department
* Attending adult poppulation

Exclusion Criteria:

* Attending exclusive maternal population

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General practitioners workin in the emergency department of hospital facilities in the Meta State.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Awareness | 30 days
  Complete identification of all items of the Alvarado score

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez Gutierrez, MD, Principal Investigator — Hospital Departamental de Villavicencio
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Result] Arroyo-Rangel C, Limon IO, Vera AG, Guardiola PM, Sanchez-Valdivieso EA. Sensitivity, Specificity and Reliability of the RIPASA Score for Diagnosis of Acute Appendicitis in Relation to the Alvarado Score. Cir Esp (Engl Ed). 2018 Mar;96(3):149-154. doi: 10.1016/j.ciresp.2017.11.013. Epub 2018 Feb 24. English, Spanish. PMID 29486897
- [Result] Sanabria-Arévalo LM, Domínguez-Torres LC, Kock J, Lotero JD, Gómez-Cáceres JC, Tuta-Quintero E. Comparison of the predictive capacity of the Alvarado and AIR scores in the diagnosis of acute appendicitis: A prospective study. Rev Gastroenterol Mex (Engl Ed). 2025;90(2):176-81.
- [Result] Caballero-Alvarado J, Rebaza-Soria S. Comparative analysis of diagnostic scales of acute appendicitis: Alvarado, RIPASA and AIR. Cir Cir. 2020;88(5):672-3.
- [Result] Bakula B, Bogut A, Karacic A, Bakula M, Maric A, Radisic Biljak V. A prospective diagnostic accuracy study of the Alvarado score in a Croatian hospital - is it time for a final conclusion? Acta Chir Belg. 2025 Aug;125(4):197-201. doi: 10.1080/00015458.2025.2512279. Epub 2025 Jun 3. PMID 40418572
- [Result] Andersson RE, Stark J. Diagnostic value of the appendicitis inflammatory response (AIR) score. A systematic review and meta-analysis. World J Emerg Surg. 2025 Feb 8;20(1):12. doi: 10.1186/s13017-025-00582-x. PMID 39923099